CLINICAL TRIAL: NCT04666025
Title: Observational Study of SARS-CoV-2 Donor-Recipient Immunity Transfer
Brief Title: SARS-CoV-2 Donor-Recipient Immunity Transfer
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20153; NCI-2020-11156 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20153 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-12-10; First posted 2020-12-14 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Accelerated Phase CML, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; Chronic Phase CML, BCR-ABL1 Positive; COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Hodgkin Lymphoma; Lymphoblastic Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; COVID-19; Hematologic Neoplasms; Hodgkin Disease; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs, blood, saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, medical chart review): DONORS: Prior to HCT, sibling donors (MRD and haplo) undergo a nasopharyngeal swab per standard of care for SARS-Cov-2 testing. For MUD donors, initial testing may consist of a questionnaire. All donors undergo collection of blood and saliva at the time of granulocyte-colony stimulating factor (G-CSF). Donors' medical charts are also reviewed.
  RECIPIENTS: Patients undergo a nasopharyngeal swab for SARS-Cov-2 testing at 30, 60, 90, 120 days post-HCT, and afterwards as deemed necessary by the treating physician. Patients also undergo the collection of blood and saliva specimens at days 30, 60, 90, 120, 150, and 180 post-HCT. Recipients' medical charts are also reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Diagnostic Laboratory Biomarker Analysis; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of nasopharyngeal swabs, blood, and saliva samples
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Electronic Health Record Review — Medical charts are reviewed
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study investigates whether donors with previous exposure to COVID-19 can pass their immunity by hematopoietic (blood) stem cell transplant (HCT) donation to patients that have not been exposed. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the virus that causes the COVID19 infection. This study may provide critical information for medical decision-making and possible immunotherapy interventions in immunocompromised transplant recipients, who are at high risk for COVID19 severe illness.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the possibility of anti-SARS-CoV-2 adaptive immunity transfer from matched related (MRD) or unrelated (MUD) HCT donor to HCT recipient.

SECONDARY OBJECTIVES:

I. To explore anti-SARS-CoV-2 adaptive immunity transfer in the haploidentical (haplo) HCT setting.

II. To assess the prevalence and change over time of SARS-CoV-2 seropositive donors among all consented donors.

OUTLINE:

DONORS: Prior to HCT, sibling donors (MRD and haplo) undergo a nasopharyngeal swab per standard of care for SARS-Cov-2 testing. For MUD donors, initial testing may consist of a questionnaire. All donors undergo collection of blood and saliva at the time of granulocyte-colony stimulating factor (G-CSF). Donors' medical charts are also reviewed.

RECIPIENTS: Patients undergo a nasopharyngeal swab for SARS-Cov-2 testing at 30, 60, 90, 120 days post-HCT, and afterwards as deemed necessary by the treating physician. Patients also undergo the collection of blood and saliva specimens at days 30, 60, 90, 120, 150, and 180 post-HCT. Recipients' medical charts are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* ALL COHORTS: Documented written informed consent of the participant
* ALL COHORTS: Recipients must have a planned allogeneic HCT procedure. MRD, MUD, and haplo HCT allowed. Usage of post-transplant cyclophosphamide (PTCy) permitted only in haplo setting
* ALL COHORTS: GCSF-mobilized peripheral blood stem cell (PBSC) only as graft source
* ALL COHORTS: Planned HCT with minimal to no-T cell depletion of graft for the treatment of the following hematologic malignancies:

  * Lymphoma (Hodgkin and non-Hodgkin)
  * Myelodysplastic syndrome
  * Acute lymphoblastic leukemia in first or second remission (for acute lymphoblastic leukemia/lymphoblastic lymphoma, the disease status must be in hematologic remission by bone marrow and peripheral blood. Persistent lymphadenopathy on computed tomography [CT] or CT/positron emission tomography [PET] scan without progression is allowed)
  * Acute myeloid leukemia in first or second remission
  * Chronic myelogenous leukemia in first chronic or accelerated phase, or in second chronic phase
  * Other hematologic malignancies including chronic lymphocytic leukemia, myeloproliferative disorders and myelofibrosis
* ALL COHORTS: Willingness to

  * Provide blood samples and saliva specimens
  * Permit medical record review
* ADDITIONAL CRITERIA FOR RECIPIENTS IN THE MAIN COHORT:

  * Absence of documented COVID-19 history and active COVID-19 infection
* ADDITIONAL CRITERIA FOR RECIPIENTS IN THE REFERENCE COHORT: Active COVID-19 infection during HCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (donors and recipients) scheduled to undergo a standard of care donor HCT procedure.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Severe acute respiratory syndrome (SARS)-Coronavirus 2 (CoV-2) Spike protein (S)-specific IgG concentration and T cell levels | Up to 180 days post-hematopoietic stem cell transplant (HCT)
  Testing for SARS-CoV-2 antibodies will be performed on serum samples using in house developed enzyme-linked immunosorbent assay (ELISA). The qualitative assays will be developed to investigate Spike subunit 1 (S1)-specific antibodies of the IgG, IgM and IgA subclasses in serum and saliva samples. All SARS-Cov-2 seropositive donor-HCT recipient pairs patients will undergo cellular immunogenicity evaluations using flow cytometry. The data analysis for estimating the effect of donor immunity transfer on functional cellular immunity through time will be exploratory in nature and will focus on graphical display and summary statistics. Longitudinal levels of T cells specific for SARS-CoV-2 S will be measured as a correlate of immunity transfer efficiency.
SARS-CoV-2 nucleocapsid protein (N) -specific IgG concentration and T cell levels | Up to 180 days post-HCT
  Testing for SARS-CoV-2 antibodies will be performed on serum samples using in house developed ELISA. The qualitative assays will be developed to investigate nucleocapsid (N)-specific antibodies of the IgG, IgM and IgA subclasses in serum and saliva samples. All SARS-Cov-2 seropositive donor-HCT recipient pairs patients will undergo cellular immunogenicity evaluations using flow cytometry. The data analysis for estimating the effect of donor immunity transfer on functional cellular immunity through time will be exploratory in nature and will focus on graphical display and summary statistics. Longitudinal levels of T cells specific for SARS-CoV-2 N antigens will be measured as a correlate of immunity transfer efficiency.
SARS-CoV-2 neutralizing antibodies | Up to 180 days post-HCT
  Evaluation of SARS-CoV-2 neutralizing antibody titers in serum samples will be performed using SARS-CoV-2 lentiviral-pseudovirus based on published protocols. Spike incorporation into the pseudovirus will be verified and quantified by western blot using Spike-specific antibodies (Sino Biological) and by ELISA using Spike Detection kit (Sino Biological), respectively.

SECONDARY OUTCOMES:
SARS-CoV-2 IgA concentration | Up to 180 days post-HCT
  Testing for SARS-CoV-2 antibodies will be performed on serum samples using in house developed ELISA.

OTHER OUTCOMES:
SARS-CoV-2 -specific T cell memory profile and associated function | Up to 180 days post-HCT
  The data analysis for estimating the effect of donor immunity transfer on functional cellular immunity through time will be exploratory in nature and will focus on graphical display and summary statistics. Longitudinal levels of T cells specific for SARS-CoV-2 S or SARS-CoV-2 N antigens will be measured as a correlate of immunity transfer efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr M Al Malki, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] La Rosa C, Chiuppesi F, Park Y, Zhou Q, Yang D, Gendzekhadze K, Ly M, Li J, Kaltcheva T, Ortega Francisco S, Gutierrez MA, Ali H, Otoukesh S, Amanam I, Salhotra A, Pullarkat VA, Aldoss I, Rosenzweig M, Aribi AM, Stein AS, Marcucci G, Dadwal SS, Nakamura R, Forman SJ, Al Malki MM, Diamond DJ. Functional SARS-CoV-2-specific T cells of donor origin in allogeneic stem cell transplant recipients of a T-cell-replete infusion: A prospective observational study. Front Immunol. 2023 Mar 3;14:1114131. doi: 10.3389/fimmu.2023.1114131. eCollection 2023. PMID 36936918
- [Derived] La Rosa C, Chiuppesi F, Park Y, Gendzekhadze K, Zhou Q, Faircloth K, Kaltcheva T, Johnson D, Ortega Francisco S, Amanam I, Otoukesh S, Pullarkat VA, Nakamura R, Diamond DJ, Forman SJ, Al Malki MM. Adoptive transfer of functional SARS-COV-2-specific immunity from donor graft to hematopoietic stem cell transplant recipients. Am J Hematol. 2022 Nov;97(11):E404-E407. doi: 10.1002/ajh.26691. Epub 2022 Sep 2. No abstract available. PMID 36053823